CLINICAL TRIAL: NCT00687947
Title: CGRP-induced Headache in Patients With Familial Hemiplegic Migraine, Migraine With Aura and Healthy Controls
Brief Title: Calcitonin Gene-related Peptide in Familial Hemiplegic Migraine (FHM) and Migraine With Aura (MA)
Acronym: CGRP-2008
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Collaborators: EUROHEAD (Other)
Responsible Party: Jakob Møller Hansen, MD, Danish Headache Center, University of Copenhagen, Faculty of Health Sciences, Department of Neurology, Glostrup Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FHM-CGRP-MA-2008
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Last update posted 2009-08-03 (Estimated); Status verified 2009-07

CONDITIONS: Familial Hemiplegic Migraine; Migraine With Aura; Healthy
Keywords: FHM; MA; healthy controls; CGRP
MeSH Terms: conditions — Migraine with Aura

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): MA-patients
  Interventions: Drug: CGRP
- 2 (Experimental): FHM-patients
  Interventions: Drug: CGRP
- 3 (Active Comparator): Healthy controls
  Interventions: Drug: CGRP

INTERVENTIONS:
Drug: CGRP — CGRP (0.5 ug/min) infused intravenously over 20 min

SUMMARY:
The aim of the present study is to explore the importance of migraine phenotype on the headache/migraine responses after CGRP in FHM-patients, MA-patients and healthy volunteers.

DETAILED DESCRIPTION:
Calcitonin gene-related peptide (CGRP) induces migraine attacks indistinguishable from spontaneous attacks in a large proportion of migraine sufferers. Treatment of spontaneous migraine attacks with an inhibitor of CGRP is effective in many patients. These data show that CGRP is involved in migraine pathophysiology.

The importance of migraine genetics is disputed. Evidence from FHM patients with known mutations indicates that migraine pathways in FHM may be different from normal migraine. The aim of the present study is to examine whether this difference also exists in FHM patients without known mutations. The project will improve our understanding of the neurobiology of migraine and stimulate development of new treatment targets.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of familial hemiplegic migraine (IHS-classification criteria)
* Diagnosis of migraine with aura(IHS-classification criteria)
* Healthy controls

Exclusion Criteria:

Patients and controls:

* A history of cerebrovascular disease and other CNS- disease
* A history of serious somatic and mental disease
* A history suggesting ischaemic heart disease
* A history of hypo- or hypertension
* Daily intake of medication apart from oral contraceptives
* Abuse of alcohol or medicine (opioid analgesics).
* Pregnant or breastfeeding women.
* On the study day:

  * No intake of a simple analgesic in the previous 48 hours
  * No headache in the previous 48 hours

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Migraine and associated symptoms | 0-14 h

SECONDARY OUTCOMES:
Migraine aura | 0 - 14 h

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Møller Hansen, MD, Principal Investigator — Danish Headache Center
Locations (1):
- Danish Headache Center, University of Copenhagen, Faculty of Health Sciences, Department of Neurology, Glostrup Hospital, Glostrup, Copenhagen, Denmark

REFERENCES:
- [Background] Hansen JM, Thomsen LL, Olesen J, Ashina M. Familial hemiplegic migraine type 1 shows no hypersensitivity to nitric oxide. Cephalalgia. 2008 May;28(5):496-505. doi: 10.1111/j.1468-2982.2008.01559.x. Epub 2008 Mar 31. PMID 18384418
- [Background] Hansen JM, Thomsen LL, Marconi R, Casari G, Olesen J, Ashina M. Familial hemiplegic migraine type 2 does not share hypersensitivity to nitric oxide with common types of migraine. Cephalalgia. 2008 Apr;28(4):367-75. doi: 10.1111/j.1468-2982.2008.01542.x. Epub 2008 Feb 22. PMID 18294248
- See also: The homepage of the Danish headache center, Glostrup, Copenhagen, Denmark — http://www.glostruphospital.dk/danishheadachecenter/menu